CLINICAL TRIAL: NCT05936840
Title: Quantitative Hormonal Biomarkers of Menstrual Health in Normal and Abnormal Cycles
Brief Title: Quantum Menstrual Health Monitoring Study
Acronym: QMHMS
Status: Recruiting | Type: Observational
Sponsor: Quanovate Tech Inc. (Industry)
Collaborators: Patricia Doyle-Baker (Unknown)
Responsible Party: Principal Investigator, Paul Yong, Associate Professor, University of British Columbia
Other Study IDs: REB23-0704
Record Dates: First submitted 2023-02-02; First posted 2023-07-10 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Menstrual Cycle Abnormal; Polycystic Ovary Syndrome; Athletes
Keywords: Quantitative urinary hormones; Follicle-stimulating hormone; Luteinizing hormone; Estrone-3-glucuronide; Pregnanediol glucuronide; Ultrasound
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Regular cycles: To characterize quantitative hormones in the urine using the Mira monitor, along with other menstrual cycle biomarkers, and validate these in reference to serum hormonal measurements and the gold-standard of the ultrasound-day of ovulation in participants with normal menstrual cycles (cycle length 24-38 days).
  Interventions: Device: Mira Monitor tracking
- Polycystic ovarian syndrome: To identify hormonal and other menstrual cycle biomarker variations in polycystic ovarian syndrome (PCOS) with oligomenorrhea.
  Interventions: Device: Mira Monitor tracking
- Athletes: To identify hormonal and other menstrual cycle biomarker variations in oligomenorrheic athletes.
  Interventions: Device: Mira Monitor tracking

INTERVENTIONS:
Device: Mira Monitor tracking — Using the Mira monitor to track the menstrual cycle

SUMMARY:
The Quantum Menstrual Health Monitoring Study will measure four key reproductive hormones in the urine to characterize patterns that predict and confirm ovulation, referenced to serum hormones and the gold-standard of the ultrasound day of ovulation in participants with regular cycles. These normal cycles will provide a reference for comparison to irregular cycles in polycystic ovarian syndrome (PCOS) and athletes. Clinical signs in the menstrual cycle (e.g. menstrual bleeding, temperature) as well as vital sign and sleep patterns will also be referenced to hormonal changes.

ELIGIBILITY:
Inclusion Criteria:

* Regularly menstruating, PCOS or athlete participants aged 18-45
* Negative pregnancy test at the beginning and at the end of each cycle
* Cycle lengths 24-34 days
* Knowledge of previous 3 cycle lengths
* Able to travel to Calgary Clinic for regular ultrasounds during the study period

Exclusion Criteria:

* For regular cycles

  * Anovulation in the last 3 cycles
  * Currently or in the previous 3 months, on medications that are known to impair or stimulate ovulation (e.g. oral contraceptives, ovulation stimulants, etc)
  * Known conditions that impair ovulation or fertility: polycystic ovarian syndrome, endometriosis, pelvic inflammatory disease in the last year, pituitary adenomas, exclusively breastfeeding
  * Previous surgeries impacting the menstrual cycle: hysterectomy, bilateral oophorectomy
  * Currently pregnant
* For PCOS and athlete groups:

  * Currently or in the previous 3 months, on medications that are known to impair or stimulate ovulation (e.g. oral contraceptives, ovulation stimulants, etc)
  * Known conditions that impair ovulation or fertility: pelvic inflammatory disease in the last year, pituitary adenomas, exclusive breastfeeding
  * Previous surgeries impacting the menstrual cycle: hysterectomy, bilateral oophorectomy
  * Currently pregnant

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Previous ultrasound studies validating urine hormone monitor measurements have targeted 50 participants over 3 cycles, for a total of 150 menstrual cycles. With 150 cycles for analysis, the study would be adequately powered to detect differences of 0.5 days in cycle parameters (with an effect size of 0.2, alpha 0.05 and power of 80%). Oversampling up to 60 participants may be required to ensure that we have 150 cycles for analysis. We will attempt to recruit 50 participants with PCOS, and 50 athletes, using the same power calculation as above.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The rise and fall of urine luteinizing hormone will predict of ovulation in all participants with confirmed ovulation | 1 year
  The LH surge on the Mira monitor will accurately predict ovulation within 1-2 days referenced to the ultrasound-day of ovulation
The rise in urine progesterone will confirm ovulation in all participants who have ovulated based on ultrasound | 1 year
  The progesterone (PDG) rise on the Mira monitor will accurately confirm ovulation within 3-5 days of the ultrasound-day of ovulation
Follicle-stimulating hormone (FSH) and estrogen (E3G) changes will predict the onset of the fertile window at least 5 days before ovulation in participants with confirmed ovulation | 1 year
  FSH and E3G changes on the Mira monitor will predict the beginning of the fertile window

SECONDARY OUTCOMES:
Menstrual bleeding scores will be correlated with changes in progesterone | 1 year
  Menstrual bleeding scores, including heavy bleeding, will be indicative of abnormal conditions like PCOS and correlated with progesterone abnormalities
Temperature rise will confirm ovulation in participants who have ovulated on ultrasound | 1 year
  Temperature, like progesterone, will rise to confirm ovulation 3-5 days after the ultrasound-confirmed day of ovulation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bouchard, MD, Study Director — University of Calgary
Locations (1):
- Thomas Bouchard, Calgary, Alberta, Canada